CLINICAL TRIAL: NCT06960161
Title: Exploring the Use of Phototherapy to Improve CPAP Compliance
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREBA.CTC-24-0059
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Phototherapy — Phototherapy

SUMMARY:
Photobiomodulation (PBM) is a type of light therapy like lasers and LEDs. PBM was previously known by different terms like "low-level laser therapy" (LLLT) or "photobiostimulation." LLLT, despite its name, can also have effects beyond biomodulation, including thermal effects useful in medical imaging and therapy.

PBM works by interacting with our biological systems, and its clinical benefits depend on factors like light wavelength, and energy output.

PBM has various clinical applications, such as wound healing, pain management, and treatment in sports injuries. It's also used as an adjunct to surgery, reducing risks and improving outcomes in areas like wound healing and inflammation. In oral medicine, PBM is applied to conditions like oral aphthous ulcers and is well-recognized for its positive effects in treatment of oral inflammation for oncology patients.

Recent studies indicate that PBM, when administered by trained professionals, can improve sleep quality and reduce snoring/SDB in adults. There's potential for its use in treating obstructive sleep apnea (OSA), showing effectiveness similar to dental sleep appliances but with fewer side effects. This effect seems to be from stabilization of the upper airway. Combining PBM with other therapies, like dental sleep appliances, has shown promise in enhancing effectiveness.

However, whether the effect of PBM in stabilizing the upper airway to reduce snoring/SDB can be used in combination with continuous positive airway pressure (CPAP) to decrease CPAP pressures and improve patient compliance has not been explored.

DETAILED DESCRIPTION:
Photobiomodulation (PBM) is a type of light therapy like lasers and LEDs. PBM was previously known by different terms like "low-level laser therapy" (LLLT) or "photobiostimulation." LLLT, despite its name, can also have effects beyond biomodulation, including thermal effects useful in medical imaging and therapy.

PBM works by interacting with our biological systems, and its clinical benefits depend on factors like light wavelength, and energy output.

PBM has various clinical applications, such as wound healing, pain management, and treatment in sports injuries. It's also used as an adjunct to surgery, reducing risks and improving outcomes in areas like wound healing and inflammation. In oral medicine, PBM is applied to conditions like oral aphthous ulcers and is well-recognized for its positive effects in treatment of oral inflammation for oncology patients.

Recent studies indicate that PBM, when administered by trained professionals, can improve sleep quality and reduce snoring/SDB in adults. There's potential for its use in treating obstructive sleep apnea (OSA), showing effectiveness similar to dental sleep appliances but with fewer side effects. This effect seems to be from stabilization of the upper airway. Combining PBM with other therapies, like dental sleep appliances, has shown promise in enhancing effectiveness.

However, whether the effect of PBM in stabilizing the upper airway to reduce snoring/SDB can be used in combination with continuous positive airway pressure (CPAP) to decrease CPAP pressures and improve patient compliance has not been explored.

ELIGIBILITY:
Inclusion Criteria:

* using CPAP
* problems with CPAP tolerance/snoring

Exclusion Criteria:

* not using CPAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
CPAP pressure | 12 months
  CPAP pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Enjoy Dental, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No